CLINICAL TRIAL: NCT02545907
Title: A Single Arm Open Labeled Multicentre Phase 1b Dose Escalation Study of Carfilzomib Taken in Combination With Thalidomide and Dexamethasone in Relapsed AL Amyloidosis
Brief Title: A Dose Escalation Study of Carfilzomib Taken With Thalidomide and Dexamethasone in Relapsed AL Amyloidosis
Acronym: CATALYST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/0786
Record Dates: First submitted 2015-08-27; First posted 2015-09-10 (Estimated); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-11

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; AL Amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — carfilzomib; Thalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KTD treatment (Experimental): Participants in the escalation phase will receive carfilzomib (K), thalidomide (T), and dexamethasone (D) in combination. The dose of thalidomide will be 50mg/day. The dose of dexamethasone will be 20mg on Day 1, 8, and 15. Carfilzomib will be administered on Day 1, 8, and 15, but the level of carfilzomib delivered with depend on the cohort allocation. The dose of carfilzomib may be:
  * Level -1 - 27mg/m2
  * Level 0 - 36mg/m2
  * Level 1 - 45mg/m2
  * Level 2 - 56mg/m2
  Participants will receive up to six cycles of treatment. Following determination of the maximum tolerated dose and recommended dose, the trial will be opened to an expansion phase where participants will receive the RD of carfilzomib, along with thalidomide and dexamethasone, using the schedule outlined above.
  Interventions: Drug: Carfilzomib; Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Lyophilized carfilzomib for injection reconstituted with water to a final concentration of 2 mg/mL.
  Other Names: Kyprolis
Drug: Thalidomide — 50mg capsule.
  Other Names: Thalidomide Celgene
Drug: Dexamethasone — 2mg tablet.
  Other Names: Decadron

SUMMARY:
This study evaluates the safety and efficacy of carfilzomib used in combination with thalidomide and dexamethasone in patients with relapsed AL amyloidosis. The trial begins with a dose escalation phase, in which the maximum tolerated and recommended dose will be determined. The trial will then open into an expansion phase in which the combination efficacy is assessed.

DETAILED DESCRIPTION:
Amyloidosis is a disorder of protein folding in which normally soluble proteins are deposited as abnormal, insoluble fibrils that progressively disrupt tissue structure and impair function. The treatment of systemic AL amyloidosis has evolved to a risk adapted approach based on the end organ damage, particularly cardiac involvement, and the functional status of the patient. Intensive therapies like high dose melphalan followed by an autologous stem cell transplant are considered for patients with limited organ involvement, younger age and excellent functional status.

The majority of patients with AL amyloidosis, however, will not be candidates for ASCT and are generally treated with combination chemotherapy. This therapy may include bortezomib, a proteasome inhibitor which is particularly effective in AL amyloidosis but which may have a severe side-effect profile.

Carfilzomib is specific for the chymotrypsin-like active site of the 20S proteasome, is structurally and mechanistically distinct from bortezomib, and has demonstrated less reactivity against non-proteasomal proteases when compared to bortezomib. It also appears to be better tolerated. However, information regarding the use of carfilzomib in the treatment of AL amyloidosis is limited.

In the dose escalation phase of this study, a minimum of 6 (3 at dose level 0 and 3 at dose level -1)and a maximum of 18 (6 at dose level 0, 1, and 2) patients will recruited in a 3+3 design with cohorts of between 3 and 6 patients, in order to determine maximum tolerated dose and recommended dose.

At the recommended dose level identified, a further 20 (minimum) patients will be recruited to further assess safety and toxicities at the RD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following characteristics are eligible for this study:

  1. Aged 18 years or greater
  2. Diagnosis of systemic AL amyloidosis with:

     * exclusion of genetic mutations associated with hereditary amyloidosis and immunohistochemical exclusion of AA and TTR amyloidosis as appropriate.
     * Amyloid related organ dysfunction or organ syndrome
  3. Measurable clonal disease
  4. Clonal relapse after previous chemotherapy or stem cell transplant OR refractory clonal disease to previous chemotherapy or stem cell transplant
  5. Capable of providing written, informed consent and willing to follow study protocol
  6. Life expectancy ≥ 6 months
  7. ECOG performance status of <3
  8. Platelet count ≥ 50x109/l)
  9. Neutrophil count ≥ 1x109/l)
  10. Haemoglobin ≥ 8g/dL
  11. Bilirubin <2 times or Alkaline phosphatase <4 times upper limit of normal.
  12. Female participants of child-bearing potential must have a negative pregnancy test prior to treatment and agree to use dual methods of contraception for the duration of the study and for 30 days following completion of study. Male participants must also agree to use a barrier method of contraception for the duration of the study and for 30 days following completion of study if sexually active with a female of child-bearing potential. Participants must comply with the Celgene pregnancy prevention programme for thalidomide

Exclusion Criteria:

* Patients with the following characteristics are ineligible for this study:

  1. Overt symptomatic multiple myeloma
  2. Amyloidosis of unknown or non AL type
  3. Localised AL amyloidosis (in which amyloid deposits are limited to a typical single organ, for example the bladder or larynx, in association with a clonal proliferative disorder within that organ)
  4. Trivial or incidental AL amyloid deposits in the absence of a significant amyloid related organ syndrome (e.g., isolated carpal tunnel syndrome).
  5. Refractory to or progressive disease with an IMid and proteasome inhibitor combination
  6. Allogeneic stem cell transplantation
  7. Solid organ transplantation
  8. Severe peripheral or autonomic neuropathy causing significant functional impairment.
  9. eGFR <20ml/min
  10. Ejection fraction < 40% or NYHA class III or IV heart failure or uncontrolled hypertension
  11. Pulmonary Hypertension
  12. Advanced Mayo stage III disease as defined by hs-Troponin T>0.07 and NT-proBNP >700 pMol/L OR NT-proBNP >1000 pMol/L OR supine SBP <100 mm of Hg
  13. Myocardial infarction in the preceeding 6 months or unstable angina or conduction abnormalities uncontrolled by medication or devices
  14. Concurrent active malignancies, except surgically removed basal cell carcinoma of the skin or other in situ carcinomas
  15. Pregnant, lactating or unwilling to use adequate contraception
  16. Systemic infection unless specific anti-infective therapy is employed.
  17. Known or suspected HIV infection
  18. Contraindication to any of the required concomitant drugs or supportive treatments. Any other clinically significant medical disease or condition or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or a participant's ability to give informed consent
  19. Previous experimental agents or approved anti-tumour treatment within 3 months before the date of registration
  20. Known allergies to the IMPs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Wechalekar, Dr, Principal Investigator — University College London, National Amyloidosis Centre
Locations (14):
- United Kingdom (14):
  - Derriford Hospital, Plymouth, Devon
  - Royal Bournemouth General Hospital, Bournemouth, Dorset
  - Guy's Hospital, London, Greater London
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - Southampton General Hospital, Southampton, Hampshire
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Birmingham Queen Elizabeth Hospital, Birmingham, West Midlands
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - St James' University Hospital, Leeds, West Yorkshire
  - Bristol Haematology and Oncology Centre, Bristol
  - The Beatson West of Scotland Cancer Centre, Glasgow

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1- Dose Level 0 - 36mg/m^2: 3 evaluable participants were recruited to dose level 0.
- Period 2 - Dose Level 1 - 45mg/m^2: 3 evaluable participants were recruited to dose level 1, one of which experienced a dose limiting toxicity.
- Period 3 - Dose Level 1 - 45mg/m^2: 4 participants were recruited to dose level 1; three of which were evaluable for the maximum tolerated dose, one of which was deemed unevaluable due experiencing an SAE after the loading dose (20 mg/m^2) of carfilzomib and was replaced.
Period: Overall Study
Arm/Group | Period 1- Dose Level 0 - 36mg/m^2 | Period 2 - Dose Level 1 - 45mg/m^2 | Period 3 - Dose Level 1 - 45mg/m^2
Started | 3 | 3 | 4
Completed | 3 | 3 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 0 - 26/mg^2; Dose Level 1 - 45/mg^2: Participants received carfilzomib (K), thalidomide (T), and dexamethasone (D) in combination. The dose of thalidomide will be 50mg/day. The dose of dexamethasone will be 20mg on Day 1, 8, and 15. Carfilzomib will be 36mg/m^2 administered on Day 1, 8, and 15,.
- Total: Total of all reporting groups
Arm/Group | Dose Level 0 - 26/mg^2 | Dose Level 1 - 45/mg^2 | Total
Number analyzed (Participants) | 3 | 7 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 6
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 75.0 [61.0 to 75.0] | 62.0 [51.0 to 73.0] | 63.0 [51.0 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities as Assessed by Reported Data
Description: Dose-Limiting Toxicities (Dose escalation phase), between the time of receiving the first registered dose of carfilzomib in cycle 1 and day 1 cycle 2, in order to establish the Maximum Tolerated Dose (MTD) of carfilzomib in combination with thalidomide and dexamethasone, will be assessed based on reported data. The number of reported dose limiting toxicities will be reported.
Time Frame: After 1 cycle of treatment; to be completed within 1 year.
Population: Evaluable set- patient who received at least one cycle of the study treatment. KTD Patients who do not receive one complete cycle due to experiencing a DLT will be included in the analysis; patients who do not receive at least one complete cycle for reasons other than toxicity, without experiencing a DLT, and who miss a dose of Carfilzomib, more than 14 doses Thalidomide or 2 doses of Dexamethasone in the first cycle, will be replaced.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 0: Participants who were allocated to receive dose level 0 and received at least one cycle of the study treatment. KTD Patients who do not receive one complete cycle due to experiencing a DLT will be included in the analysis; patients who do not receive at least one complete cycle for reasons other than toxicity, without experiencing a DLT, and who miss a dose of Carfilzomib, more than 14 doses Thalidomide or 2 doses of Dexamethasone in the first cycle, will be replaced.
- Dose Level 1: Participants who were allocated to receive dose level 1 and received at least one cycle of the study treatment. KTD Patients who do not receive one complete cycle due to experiencing a DLT will be included in the analysis; patients who do not receive at least one complete cycle for reasons other than toxicity, without experiencing a DLT, and who miss a dose of Carfilzomib, more than 14 doses Thalidomide or 2 doses of Dexamethasone in the first cycle, will be replaced.
Arm/Group | Dose Level 0 | Dose Level 1
Number analyzed (Participants) | 3 | 6
Participants | 0 | 1

2. Primary Outcome: Number of Participants Experiencing Grade 3 or 4 Toxicity as Assessed by CTCAE v4.0.
Description: The percentage of patients treated who experience any grade 3 or 4 toxicity as assessed by CTCAE v4.0 throughout all treatment cycles will be assessed based on reported data.
Time Frame: Between informed consent provided and 30 days post last trial treatment administration, up to 7 months
Population: All patients that receive at least one dose of Carfilzomib and with no protocol deviations with relevant impact on safety will be included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 0- Safety Population: All patients allocated to dose level 0 that received at least one dose of Carfilzomib and with no protocol deviations with relevant impact on safety will be included in the safety analysis set.
- Dose Level 1- Safety Population: All patients allocated to dose level 1 that received at least one dose of Carfilzomib and with no protocol deviations with relevant impact on safety will be included in the safety analysis set.
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants | 2 | 3

3. Secondary Outcome: Clonal Response Rate Within 3 Months, at 3 Months, Within 6 Months and at 6 Months as Determined by Paraprotein and Free Light Chain Assessment.
Description: Participant clonal response rate within 3 months, at 3 months, within 6 months and at 6 months will be assessed. The percentage of participants who achieve at least a partial response will be reported.
  Clonal response is defined as:
  CR: Negative immunofixation of serum and urine (serum alone in anuric patients) AND normal FLC concentration and kappa/lambda FLC ratio (FLC ratio alone in renal failure) AND ≤5% plasma cells in bone marrow without clonality by immunohistochemistry or immunofluorescencea
  VGPR: >90% reduction in serum paraprotein or abnormal component of FLC or dFLC over the starting value or dFLC <40mg/L
  PR: ≥50% decrease in aberrant FLC concentration or dFLC (or ≥50% decrease in dFLC if renal failure) or serum paraprotein but not fulfilling criteria for CR or VGPR
  MR: >25% but <50% decrease in aberrant FLC or dFLC or paraprotein
  NR: Not meeting FLC criteria for CR, PR or MR
Time Frame: Within 3 months, at 3 months, within 6 months and at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants
  Within 3 cycles | 1 | 5
  At the end of cycle 3 | 1 | 5
  Within 6 cycles | 2 | 5
  At the end of cycle 6 | 2 | 5

4. Secondary Outcome: Amyloidotic Organ Response Rate Within 3 Months and 6 Months Based on Biochemical, Electrocardiographical, and Radiographical Assessment.
Description: Amyloidotic organ response rate is assessed using the following criteria:
  Heart - Interventricular septal thickness decreased by 2 mm or 10% improvement in ejection fraction or a 30% and 35 pMol/L reduction in NT-ProBNP (only applicable if there is no change or <25% improvement in renal function) or significant improvement in lateral wall TDI S wave and E/E' ratio
  Kidney - 50% decrease (at least 0.5 g/day) in 24-hr urinary protein loss (urine protein must be>0.5 g/day pretreatment) without fall in creatinine clearance of ≥25% from baseline
  Liver - 50% decrease in abnormal alkaline phosphatase value or a decrease in liver size radiographically by at least 2 cm
  Nerve - Improvement in electromyogram nerve conduction velocity
  Soft tissue - Definite clinical and/or radiographic improvement with associated functional improvement in affected tissue.
  The percentage of patients who achieve organ response within 3 and 6 months of trial registration will be reported.
Time Frame: Within 3 months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants
  Response within 3 months | 0 | 0
  Response within 6 months | 0 | 0
  No response | 3 | 7

5. Secondary Outcome: Time to Amyloidotic Organ Response Based on Reported Data.
Description: The time to amyloidotic organ response (as outlined above) will be assessed based on reported data. The number of months this takes will be reported.
Time Frame: Within 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants | 0 | 0

6. Secondary Outcome: Number of Deaths at 6 Months Based on Reported Data.
Description: The number of deaths at 6 months will be assessed and reported based on reported data.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants | 0 | 0

7. Secondary Outcome: Number of Patients Progression-free at 6 Months Based on Reported Data.
Description: The number of patients who are progression-free at 6 months will be assessed based on reported data. Patients who are progression-free will have not had an haematological relapse or organ progression.
  Haematological relapse is defined as:
  From CR: Increase in the aberrant serum free light chain concentration to outside the normal range and by a factor of ≥2 from that at the time of CR or re-appearance of the original paraprotein
  From PR or VGPR: Increase in the aberrant free light chain concentration by a factor of ≥2 from that at the time of PR (≥50% change in ratio away from normal in patients with renal failure) or doubling of the serum paraprotein level (if starting >5g/L) or doubling and increase of serum paraprotein to >5g/L (if starting <5g/L)
  Organ progression is defined, by organ, as:
  Heart: Interventricular septal thickness increased by >2 mm compared with baseline or 20% decline in ejection fraction
  Kidney: 50% increase (at least 1 g/day) in 24-hr urinary
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants | 3 | 7

8. Secondary Outcome: Maximum Response Determined by Paraprotein and Free Light Chain Assessment.
Description: The maximum response to therapy will be determined by assessing the best reported response for each participant. Maximum response will be determined based on free light chain and paraprotein assessments by the National Amyloidosis Centre. The data will be reported using the response rates observed (complete, very good partial, partial, no response).
Time Frame: Within 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants
  No response | 1 | 0
  Partial response | 0 | 1
  Very good partial response | 2 | 1
  Complete response | 0 | 3
  Not evaluable | 0 | 2

9. Secondary Outcome: Time to Maximum Response Based on Reported Data.
Description: The time to maximum response to treatment will be assessed by determining the time required for each participant to achieve maximum response (defined above), and will be presented on Kaplan-Meier curves. The number of months taken to achieve this maximum response will be reported. Time to maximum response was analysed overall only, and not by arm due the small sample size.
Time Frame: Within 6 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Safety Population: All patients that received at least one dose of Carfilzomib and with no protocol deviations with relevant impact on safety will be included in the safety analysis set..
Arm/Group | Safety Population
Number analyzed (Participants) | 10
months | 5.3 [NA to NA] — Seven out of 10 participants achieved a maximum response. Two participants who experienced DLTs were not evaluable for response and one participant who discontinued after two cycles of treatment did not achieve a response. Corresponding 95% confidence intervals is not calculable due to the low number of events.

10. Secondary Outcome: Number of Patients Withdrawing From Treatment Based on Reported Data.
Description: The number of patients withdrawing from treatment will be assessed based on reported data.
Time Frame: Within 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants | 0 | 0

11. Secondary Outcome: Number of Patients Experiencing Dose Delays Based on Reported Data.
Description: The number of patients experiencing dose delays will be assessed based on reported data.
Time Frame: Within 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants | 2 | 1

12. Secondary Outcome: Compliance Profile of KTD Based on Reported Chemotherapy Compliance Data.
Description: The compliant profile of participants to KTD will be assessed by determining the number of missed doses from recorded data. Participants will be regarded as compliant if participants have missed no more than 14 days of thalidomide, 2 days of dexamethasone, and 1 dose of carfilzomib per cycle. Compliance will be reported in terms of the number of participants who were compliant.
Time Frame: Within 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0- Safety Population | Dose Level 1- Safety Population
Number analyzed (Participants) | 3 | 7
Participants | 1 | 5

ADVERSE EVENTS:
Time Frame: All adverse events that occur between informed consent and 30 days post last trial treatment administration must be recorded in the patient notes and the trial CRFs, up to 7 months.
Description: Definitions are the same as those in clinicialtrials.gov
Groups:
- Dose Level 0 - Safety Population: All patients allocated to dose level 0 that received at least one dose of Carfilzomib and with no protocol deviations with relevant impact on safety will be included in the safety analysis set.
- Dose Level 1 - Safety Population: All patients allocated to dose level 1 that received at least one dose of Carfilzomib and with no protocol deviations with relevant impact on safety will be included in the safety analysis set.
Arm/Group | Dose Level 0 - Safety Population | Dose Level 1 - Safety Population
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/7
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 - Safety Population (N=3) | Dose Level 1 - Safety Population (N=7)
Abdominal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury on CKD (Investigations) | 0 (0) | 1 (1)
Fever (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 - Safety Population (N=3) | Dose Level 1 - Safety Population (N=7)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Social circumstances - Other, specify (Social circumstances) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 5 (5)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Ggt Increased (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 1 (1)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bladder Infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial closed to recruitment following the dose escalation stage without opening the expansion phase due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT02545907/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02545907/SAP_001.pdf